CLINICAL TRIAL: NCT04395456
Title: A Phase 2 Clinical Trial to Assess the Safety and Efficacy of Complement 3 Inhibitor, AMY-101, in Patients With Acute Respiratory Distress Syndrome Due to COVID-19 (SAVE)
Brief Title: A Study of the C3 Inhibitor AMY-101 in Patients With ARDS Due to COVID-19 (SAVE)
Acronym: SAVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amyndas Pharmaceuticals S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMY-101_SAVE
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Acute Respiratory Distress Syndrome Due to SARS-CoV-2 Infection (Severe COVID19)
MeSH Terms: conditions — COVID-19 | interventions — AMY-101; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMY-101 (Experimental)
  Interventions: Drug: AMY-101
- Placebo (Placebo Comparator)
  Interventions: Other: WFI 5% glucose

INTERVENTIONS:
Drug: AMY-101 — C3 complement inhibitor
  Arms: AMY-101
Other: WFI 5% glucose — Placebo
  Arms: Placebo

SUMMARY:
The study is a prospective, randomized, placebo-controlled, single-blind phase 2 clinical study of the efficacy and safety of AMY-101, a potent C3 inhibitor, for the management of patients with ARDS caused by SARS-CoV-2 infection.

We will assess the efficacy and safety, as well as pharmacokinetics (PK), and pharmacodynamics (PD). The study will assess the impact of AMY-101 in patients with severe COVID19; specifically, it will assess the impact of AMY-101 1) on survival without ARDS and without oxygen requirement at day 21 and 2) on the clinical status of the patients at day 21.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Acute Respiratory Distress Syndrome due to SARS-CoV-2 infection (severe Covid-19), according to the following criteria:

  1. Demonstration of SARS-CoV-2 RNAemia in nasopharyngeal swap or bronchio-alveolar lavage (BAL)
  2. A ratio of the partial pressure of oxygen (PaO2) to the fraction of inspired oxygen (FiO2), PaO2/FIO2, ≤300 mmHg

     * Mild ARDS (PaO2/FIO2, ≤300 and >200 mm Hg);
     * Moderate ARDS (PaO2/FIO2, ≤200 and >100 mm Hg);
     * Severe ARDS (PaO2/FIO2, ≤100 mm Hg);
  3. Pulmonary infiltrates suggestive of SARS-COV-2-related ARDS: e.g., bilateral infiltrates at chest X-ray or B-lines at lung US scan.
* Dated and signed informed consent from patient or legal represantative.

Exclusion Criteria:

* Intubated patients
* Demonstrated or suspected uncontrolled systemic severe infection, such as sepsis (e.g.: positive blood culture, or procalcitonin ≥0.25 µg/L)
* Demonstrated local extrapulmonary abscess
* ARDS due to cardiac failure or fluid overload
* Concomitant treatment with immunomodulatory /immunosuppressive drugs , which have potential activity against the disease
* Multi Organ Failure (MOF)
* Severe renal failure (CKD, by defition glomerular filtration rate <30 ml/min)
* Neisseria meningitidis infection that is not resolved
* Current treatment with a complement inhibitor
* Intravenous immunoglobulin (IVIg) within 3 weeks prior to Screening
* Participation in another interventional treatment study within 30 days before initiation of the study treatment (Day 1 in this study) or within 5 half-lives of that investigational product, whichever is greater.
* Chemotherapy for less than 3months
* Pregnancy
* Age <18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who are alive, without evidence of ARDS (i.e. PaO2/FIO2 >300 mm Hg), who do not require any oxygen support (in room air). | 21 days
The proportion of patients assigned to each category, of a six-category ordinal scale. | 21 days
  The clinical status is based on the following six-category ordinal scale:
  * 1: not hospitalised;
  * 2: hospitalised, not requiring supplemental oxygen;
  * 3: hospitalised, requiring supplemental oxygen;
  * 4: hospitalised, requiring nasal high-flow oxygen therapy, non-invasive mechanical ventilation, or both;
  * 5: hospitalised, requiring ECMO, invasive mechanical ventilation, or both; and
  * 6: death.

SECONDARY OUTCOMES:
The proportion of patients assigned to each category, of a six-category ordinal scale. | On days 7, 14, and 44
  The clinical status is based on the following six-category ordinal scale:
  * 1: not hospitalised;
  * 2: hospitalised, not requiring supplemental oxygen;
  * 3: hospitalised, requiring supplemental oxygen;
  * 4: hospitalised, requiring nasal high-flow oxygen therapy, non-invasive mechanical ventilation, or both;
  * 5: hospitalised, requiring ECMO, invasive mechanical ventilation, or both; and
  * 6: death.
Proportion of patients surviving | Through to day 44
Proportion of respiratory failure-free survival | Day 44
  With respiratory failure defined as any of the following:
  1. Worsening of severe gas transfer deficit, accounting for a shift in ARDS disease category (PaO2/FiO2 ≤200 for patients with PaO2/FiO2 >200 at baseline; PaO2/FiO2 ≤100 for patients with PaO2/FiO2 >100 at baseline),
  2. Persistent respiratory distress while receiving oxygen (persistent marked dyspnea,use of accessory respiratory muscles, paradoxical respiratory movements),
  3. Transfer to the intensive care unit for intubation,
  4. Death.
Cumulative incidence of resolution of ARDS (defined as PaO2/FiO2 ≥200 in room air) | Through day 44
Cumulative incidence of freedom from oxygen requirement | Through day 44
Proportion of patients requiring invasive mechanical ventilation due to worsening of ARDS | Within 14 days after inclusion in the study
Proportion of patients requiring non-invasive mechanical ventilation (NIV) due to worsening of ARDS | Within 14 days after inclusion in the study
Proportion of patients developing thrombotic microangiopathies | Through day 44
Changes in PaO2 and PaO2/FIO2 | Through day 44
Changes in quick Sequential Organ Failure Assessment Score (qSOFA: respiratory rate, systolic blood pressure, Glasgow Coma Scale (GCS) | Through day 44
Changes in maximal and minimal cardiovascular parameters: Respiratory rate | Through day 44
Changes in maximal and minimal cardiovascular parameters: Heart Rate | Through day 44
Changes in levels of biomarkers of inflammation (CBC, CRP, Ferritin, Procalcitonin, D-dimers, LDH) | On days 0, 1, 2, 4, 7, 10, 14, 21 and 44
Length of stay in ICU | Through day 44
Cumulative incidence of discharge from hospital | Through day 44
Number of adverse events | Through day 44
Changes in levels of anti-drug antibodies | On day 0 , 14 and 44
Changes in levels of biomarkers of complement activity: C3, C3a, C5a, sC5b-9 | On days 0, 1, 2, 4, 7, 10, 14, 21 and 44
Changes in levels of biomarkers of cytokine release syndrome: IL-1, IL-6, IL-12 | On days 0, 1, 2, 4, 7, 10, 14, 21 and 44
Changes in levels of Club Cell protein CC16 (biomarker of lung damage ) | On days 0, 1, 2, 4, 7, 10, 14, 21 and 44
Changes in levels of AMY-101 plasma level | On days 1, 2, 4, 7, 10, 14, 15, 21

REFERENCES:
- [Background] Risitano AM, Mastellos DC, Huber-Lang M, Yancopoulou D, Garlanda C, Ciceri F, Lambris JD. Complement as a target in COVID-19? Nat Rev Immunol. 2020 Jun;20(6):343-344. doi: 10.1038/s41577-020-0320-7. Epub 2020 Apr 23. PMID 32327719
- [Background] Mastaglio S, Ruggeri A, Risitano AM, Angelillo P, Yancopoulou D, Mastellos DC, Huber-Lang M, Piemontese S, Assanelli A, Garlanda C, Lambris JD, Ciceri F. The first case of COVID-19 treated with the complement C3 inhibitor AMY-101. Clin Immunol. 2020 Jun;215:108450. doi: 10.1016/j.clim.2020.108450. Epub 2020 Apr 29. PMID 32360516